CLINICAL TRIAL: NCT00746226
Title: Probiotic Intervention for Children With Birch Pollen Allergy
Brief Title: Probiotics for Birch Pollen Allergy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Danisco (Industry)
Responsible Party: E. Isolauri Professor, Turku University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Danisco - TBPA06
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2008-09-03 (Estimated); Status verified 2008-09

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: birch pollen
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Numbers 509-513, 700-709 and 900-909 Probiotic combination of L. acidophilus and B. lactis
  Interventions: Biological: Lactobacillus acidophilus and Bifidobacterium lactis
- B (Placebo Comparator): Numbers 612-624 and 800-811
  Microcrystalline cellulose
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lactobacillus acidophilus and Bifidobacterium lactis — Daily 5x10^9 CFU of a combination of L. acidophilus and B. lactis
  Arms: A
Biological: Placebo — Microcrystalline cellulose
  As capsule which could be opened
  Arms: B

SUMMARY:
Birch pollen allergy is one of the most common forms of respiratory allergy in the Nordic countries. Treatment consists of antihistamine use. Specific probiotic strains have been observed to modulate the immune system. Since the body has a common mucosal immune system; it was hypothesised that consumption of probiotics may affect also the respiratory mucosal immune response and hence affect respiratory allergy.

Earlier studies with probiotics had been unable to show improvements in adults with pollen allergy. It was therefore hypothesised that children, who's immune system is not yet fully developed, might be better targets.

ELIGIBILITY:
Inclusion Criteria:

Physician verified birch pollen allergy

Exclusion Criteria:

Diagnosed asthma Habitual use of probiotics and/or prebiotics

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2006-03; Primary Completion 2006-06 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Birch pollen allergy symptoms | March/April and June
Nasal Eosinophilia | April/May and June

SECONDARY OUTCOMES:
Change in microbiota composition | April/May and June
Cytokine profile from serum | April/May and June
Faecal recovery of administered probiotics | April/May and June

CONTACTS AND LOCATIONS:
Overall Officials: Arthur C Ouwehand, PhD, Study Chair — Danisco
Locations (1):
- Turku University Central Hospital, Turku, Finland